CLINICAL TRIAL: NCT04668638
Title: Impact of Respiratory Rehabilitation on Quality of Life, Measures by the SF-36 Score, in Patients With Hyperventilation Syndrome: Crossover, Prospective and Randomized Study
Brief Title: Impact of Respiratory Rehabilitation on Quality of Life in Patients With Hyperventilation Syndrome
Acronym: RESPIR-HVS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHRO-2020-19
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hyperventilation Syndrome
Keywords: Hyperventilation syndrome; Respiratory rehabilitation; Quality of Life

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two groups:
  * Group 1 (Control Group) will not immediately receive respiratory rehabilitation but between the 2nd and 4th months postdiagnosis.
  * Group 2 (Intervention Group) will immediately receive rehabilitation between the diagnosis and the 2nd month postdiagnosis.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Group 1 (Control Group) will not immediately receive respiratory rehabilitation but between the 2nd and 4th months postdiagnosis.
  Interventions: Other: Respiratory rehabilitation
- Intervention group (Other): Group 2 (Intervention Group) will immediately receive rehabilitation between the diagnosis and the 2nd month postdiagnosis.
  Interventions: Other: Respiratory rehabilitation

INTERVENTIONS:
Other: Respiratory rehabilitation — Respiratory rehabilitation includes education, hypoventilation exercises, diaphragmatic breathing exercises, relaxation, retraining, others.

SUMMARY:
The hyperventilation syndrome is a quite frequent pathology, affecting up to 10% of the general population and 40% of the asthmatic population. Its physiopathology is still badly known and even if it is a benign affection, its associated comorbidities and symptomatology greatly decrease the patients' quality of life. Yet, no medicinal treatments have been proved useful, but prescribers noticed improvements after physiotherapy. Given that the physiotherapy impact on hyperventilation syndrome is not well described in the literature, this study aims to scientifically ascertain physiotherapy benefits on quality of life and symptomatology in hyperventilation syndrome-suffering patients.

ELIGIBILITY:
Inclusion Criteria:

* Positive hyperventilation syndrome diagnosis
* Having a social security insurance
* Being at least 18 years old
* Having given their written consent

Exclusion Criteria:

* Being put under guardianship or curatorship
* Having seen a physiotherapist for a respiratory rehabilitation in the last three months
* Suffering from a chronic and degenerative pathology (chronic obstructive pulmonary disease, Parkinson's disease, idiopathic fibrosis, …)
* Not being able to receive the respiratory rehabilitation from our care providers
* Already having received a rehabilitation for hyperventilation syndrome
* Not speaking French or not being unable to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Incidence of respiratory rehabilitation on Quality of life | Day 0
  Quality of life will be evaluated with the SF-36 score
Incidence of respiratory rehabilitation on Quality of life | Month 2
  Quality of life will be evaluated with the SF-36 score
Incidence of respiratory rehabilitation on Quality of life | Month 4
  Quality of life will be evaluated with the SF-36 score

SECONDARY OUTCOMES:
Change in symptomatology | Day 0
  Change in symptomatology will be evaluated on the Nijmegen questionnaire
Change in symptomatology | Month 2
  Change in symptomatology will be evaluated on the Nijmegen questionnaire
Change in symptomatology | Month 4
  Change in symptomatology will be evaluated on the Nijmegen questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Louis-François BIRNESSER, Principal Investigator — CHR Orléans
Locations (1):
- CHR d'Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gardner WN. The pathophysiology of hyperventilation disorders. Chest. 1996 Feb;109(2):516-34. doi: 10.1378/chest.109.2.516. No abstract available. PMID 8620731
- [Background] Lewis RA, Howell JB. Definition of the hyperventilation syndrome. Bull Eur Physiopathol Respir. 1986 Mar-Apr;22(2):201-5. PMID 3708188
- [Background] Thomas M, McKinley RK, Freeman E, Foy C. Prevalence of dysfunctional breathing in patients treated for asthma in primary care: cross sectional survey. BMJ. 2001 May 5;322(7294):1098-100. doi: 10.1136/bmj.322.7294.1098. PMID 11337441
- [Background] Lewis T, Cotton, Barcroft J, Dufton D, Milroy TR, Parsons TR. BREATHLESSNESS IN SOLDIERS SUFFERING FROM IRRITABLE HEART. Br Med J. 1916 Oct 14;2(2911):517-9. doi: 10.1136/bmj.2.2911.517. No abstract available. PMID 20768329
- [Background] van Dixhoorn J, Duivenvoorden HJ. Efficacy of Nijmegen Questionnaire in recognition of the hyperventilation syndrome. J Psychosom Res. 1985;29(2):199-206. doi: 10.1016/0022-3999(85)90042-x. PMID 4009520
- [Background] Vansteenkiste J, Rochette F, Demedts M. Diagnostic tests of hyperventilation syndrome. Eur Respir J. 1991 Apr;4(4):393-9. PMID 1855568
- [Background] Nixon PG. Effort syndrome: hyperventilation and reduction of anaerobic threshold. Biofeedback Self Regul. 1994 Jun;19(2):155-69. doi: 10.1007/BF01776488. PMID 7918753
- [Background] Chenivesse C, Similowski T, Bautin N, Fournier C, Robin S, Wallaert B, Perez T. Severely impaired health-related quality of life in chronic hyperventilation patients: exploratory data. Respir Med. 2014 Mar;108(3):517-23. doi: 10.1016/j.rmed.2013.10.024. Epub 2013 Nov 7. PMID 24269004
- [Background] Kraft AR, Hoogduin CA. The hyperventilation syndrome. A pilot study on the effectiveness of treatment. Br J Psychiatry. 1984 Nov;145:538-42. doi: 10.1192/bjp.145.5.538. PMID 6388711
- [Background] Van De Ven LL, Mouthaan BJ, Hoes MJ. Treatment of the hyperventilation syndrome with bisoprolol: a placebo-controlled clinical trial. J Psychosom Res. 1995 Nov;39(8):1007-13. doi: 10.1016/0022-3999(95)00508-0. PMID 8926595
- [Background] Hoes MJ, Colla P, Folgering H. Clomipramine treatment of hyperventilation syndrome. Pharmakopsychiatr Neuropsychopharmakol. 1980 Jan;13(1):25-8. doi: 10.1055/s-2007-1019606. PMID 7367465
- [Background] Jones M, Harvey A, Marston L, O'Connell NE. Breathing exercises for dysfunctional breathing/hyperventilation syndrome in adults. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD009041. doi: 10.1002/14651858.CD009041.pub2. PMID 23728685